CLINICAL TRIAL: NCT03367143
Title: A Phase II Study of the Efficacy and Safety of Lenalidomide Plus ICE in the Treatment of Refractory and Relapsed Diffuse Large B-cell Lymphoma
Brief Title: Lenalidomide Plus ICE in the Treatment of Refractory and Relapsed DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-ICE
Record Dates: First submitted 2017-11-10; First posted 2017-12-08 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Diffuse Large B-Cell Lymphoma Refractory
MeSH Terms: interventions — Lenalidomide; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-ICE (Experimental): Lenalidomide 25mg/d po d1-10, Ifosfamide 1500mg/m2/d iv d1-3, Carboplatin 5*[GFR(ml/min)+25]mg/d iv d2, Etoposide 100mg/m2/d iv d1-3, Frequency every 21 days, Total cycles 4
  Interventions: Drug: Lenalidomide; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Lenalidomide
Drug: Ifosfamide
Drug: Carboplatin
Drug: Etoposide

SUMMARY:
This study is to evaluate the efficacy and safety of Lenalidomide plus ICE in the treatment of Refractory and Relapsed DLBCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diffuse large B-cell lymphoma. Previously treated with 1, and only 1, chemotherapy regimen including rituximab and anthracycline. Relapse after CR, less than PR or PR to previous treatment.
2. No history of stem cell transplantation.
3. Age between 16-75.
4. ECOG<3.
5. At least 1 measurable tumor mass.
6. Minimum life expectancy of 3 months.
7. Written informed consent.
8. No history of using Lenalidomide, ifosfamide, carboplatin and etoposide.
9. No uncontrolled CNS involvement by lymphoma:No CNS disease at time of relapse;CNS disease diagnosed at initial presentation allowed provided a complete response for CNS disease was achieved and maintained.

Exclusion Criteria:

1. Chemotherapy or large field radiotherapy within 3 weeks prior to entering the study.
2. Clinically significant active infection.
3. Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule.
4. Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.
5. Subject has ≥grade 2 peripheral neuropathy or grade 1 with pain within 14 days before enrollment.
6. Patients who are pregnant or breast-feeding.
7. HIV infection.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 12 weeks

SECONDARY OUTCOMES:
Progression free survival rate | 1 year
Overall survival rate | 1 year
Overall response rate | 12 weeks
Safety as assessed using CTCAE v4.0 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No